CLINICAL TRIAL: NCT02373826
Title: Novel Method for Real Time Co-Registration of IVUS and Coronary Angiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0028-13-HYMC
Record Dates: First submitted 2015-02-16; First posted 2015-02-27 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Intravascular Ultrasound (IVUS) Angiography Co-registration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
During coronary angiography, the lumen of the arteries is imaged but intravascular ultrasound (IVUS) is necessary to determine the plaque extension and its composition, lesion length and luminal reference diameter. We aimed to investigate the accuracy, feasibility, safety and value of a novel method for co-registration of IVUS and coronary angiographic images.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine coronary angioplasty

Exclusion Criteria:

* Cardiogenic shock
* Acute myocardial infarction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine coronary angioplasty
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Co-Registration of IVUS and Coronary Angiography | One month
  For determination of the accuracy of the co-registration feature, and the accuracy and precision of the length measurements, a flexible phantom was used in order to simulate an artery and enable simulation of the cardiac motion. The sample size for testing the co-registration algorithm was 108 samples (each sample was defined as a landmark). The resultant mean of the absolute distance accuracy was 0.995 mm with a standard deviation of 0.809 mm. The statistical validation in phantoms, resulted in an accuracy of 1.12 mm, meeting the original specification.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel